CLINICAL TRIAL: NCT06461767
Title: Repetitive Transcranial Magnetic Stimulation in Treatment of Chronic Migraine
Brief Title: Repetitive Transcranial Magnetic Stimulation in Treatment and Prophylaxis of Chronic Migraine in Patients With no Prophylactic Treatment for the Last 3 Months
Acronym: rTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tarik Mohamed Abdelnaeem, principal investigator, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-05-06MS
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Intervention Model Description: the patient will divide into 4 groups first group will receive stimulation over the left motor cortex second group will receive stimulation over left dorsolateral prefrontal cortex third group will receive stimulation over both left motor cortex and left dorsolateral prefrontal cortex fourth group will receive sham stimulation
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group (1) will rTMS over left motor cortex (Active Comparator): Repetitive transcranial magnetic stimulation parameters:
  stimulation site: left motor cortex intensity: 70% of resting motor threshold frequency: 15 Hz number of pulses: 30 number of trains: 40
  Interventions: Device: transcranial magnetic stimulation device
- group (2) will receive rTMS over left dorsolateral prefrontal cortex (Active Comparator): Repetitive transcranial magnetic stimulation parameters:
  stimulation site: left dorsolateral prefrontal cortex intensity: 70% of resting motor threshold frequency: 15 Hz number of pulses: 30 number of trains: 40
  Interventions: Device: transcranial magnetic stimulation device
- group (3) will receive rTMS over left dorsolateral prefrontal cortex and left motor cortex (Active Comparator): Repetitive transcranial magnetic stimulation parameters:
  stimulation site: left dorsolateral prefrontal cortex and left motor cortex intensity: 70% of resting motor threshold frequency: 15 Hz number of pulses: 30 number of trains: 40
  Interventions: Device: transcranial magnetic stimulation device
- group (4) will receive sham stimulation (Sham Comparator): Repetitive transcranial magnetic stimulation parameters:
  stimulation site: the coil will be perpendicular over vertex of skull intensity: 70% of resting motor threshold frequency: 15 Hz number of pulses: 30 number of trains: 40
  Interventions: Device: transcranial magnetic stimulation device

INTERVENTIONS:
Device: transcranial magnetic stimulation device — Repetitive transcranial magnetic stimulation parameters:
  stimulation site: left dorsolateral prefrontal cortex and left motor cortex intensity: 70% of resting motor threshold frequency: 15 Hz number of pulses: 30

SUMMARY:
Compared with the patients with episodic migraine those with chronic migraine have worst quality of life and more severe headache related disability we investigate Repetitive transcranial magnetic stimulation in treatment and prophylaxis of chronic migraine

ELIGIBILITY:
Inclusion criteria:

* A study sample of patients with chronic migraine according to international classification of headache disorders-3 (ICHD-3).
* Patients are regular on follow up visits.

Exclusion criteria:

* Patients with depression by Hamiliton scale of depression by using its Arabic version Translated by Dr Lotfy Fateem
* patients on prophylactic medications for chronic migraine.
* pregnancy.
* cochlear implants, cardiac pacemaker, and metal body implanted in head-and-neck region.
* Patients refused to give informed consent.
* History of seizures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
improvement of headache severity and number of attacks of headache before and after intervention by visual analogue scale and headache impact test | one month after treatment
  improvement of headache severity and number of attacks of headache before and after intervention by visual analogue scale and headache impact test

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mohamed, Principal Investigator — Sohag faculty of medicine
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR